CLINICAL TRIAL: NCT00462631
Title: Paclitaxel-Eluting Balloon Angioplasty and Cobalt-Chromium Stents Versus Conventional Angioplasty and Paclitaxel-Eluting Stents in the Treatment of Native Coronary Artery Stenoses of Diabetic Patients
Brief Title: Paclitaxel Eluting Balloon Versus Drug Eluting Stent in Native Coronary Artery Stenoses of Diabetic Patients
Acronym: PEPCAD IV
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Heart Centre Rotenburg (Other)
Collaborators: B. Braun Medical SA (Industry)
Responsible Party: Principal Investigator, Ralf Degenhardt, PhD, Data Manager, Heart Centre Rotenburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBM-VS-55; PEPCAD IV/CRI/06-03/n-c
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Stenosis; Diabetes Mellitus
Keywords: coronary artery; Diabetes
MeSH Terms: conditions — Coronary Stenosis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): paclitaxel eluting balloon followed by bare metal stent
  Interventions: Device: Paclitaxel Eluting Balloon; Device: bare metal stent
- 2 (Active Comparator): Paclitaxel eluting stent
  Interventions: Device: paclitaxel eluting stent

INTERVENTIONS:
Device: Paclitaxel Eluting Balloon — Paclitaxel eluting balloon
  Arms: 1
Device: paclitaxel eluting stent — paclitaxel eluting stent
  Arms: 2
Device: bare metal stent — bare metal stent
  Arms: 1

SUMMARY:
The aim of the study is to compare the efficacy of Paclitaxel-eluting PTCA-balloon dilation (SeQuentTM Please) followed by cobalt-chromium stent (CoroflexTM Blue) deployment versus Paclitaxel-eluting stent (TaxusTM LibertéTM) deployment in the treatment of de-novo-stenoses in native coronary arteries (reference diameter:more then 2.5 mm and below 3.5 mm, length of stenosis ≥ 10 mm ≤ 20 mm) of patients with diabetes mellitus for ≥ 3 years for procedural success and preservation of vessel patency.

This study is a prospective, randomized, multi-center, two-armed phase-II pilot study conducted in Malaysia and Thailand.

128 diabetes mellitus patients shall complete the study per protocol after random assignment to either of the treatment groups on the order of 20 to 50 patients per center.

Diabetes mellitus patients with stable or selected forms of unstable angina or documented ischemia due to a de-novo stenosis in a native coronary artery will be enrolled. Vessels may not supply an entirely infarcted myocardial area.

Late lumen loss at 9 months is the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* History of diabetes mellitus of at least 3 yrs prior to enrollment. Diabetes mellitus may be treated either orally or s.c.
* Stable blood glucose level for the 6 months preceding enrollment as reflected by HbA1c concentrations measured exclusively ≤ 8 %
* Patients with stable angina pectoris (CCS class 1-3) or with unstable angina pectoris (Braunwald class 1-2, A-C) or documented ischemia or with documented silent ischemia
* Patients eligible for coronary revascularization by means of PCI
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 6 months follow-up
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 9 months angiographic follow-up
* Patients must agree to undergo the 3 year clinical follow-up
* De-novo native coronary artery stenosis (reference diameter: ≥2.5 mm and ≤ 3.5 mm, length of stenosis: ≥ 10 mm and ≤ 20 mm)
* Target lesion is ≥ 3 mm distant from a major side branch (> 2.0 mm in diameter) and ≥ 3 mm form a previously deployed stent of any type (including active and passive coatings, bare metal stents)
* The target lesion must be treated with a single stent only (multiple stenting shifts the patient to the intention-to-treat group)
* Single or multi-vessel coronary artery disease

Exclusion Criteria:

* Patients with acute (< 24 h) or recent (48 hours) myocardial infarction
* Patients with unstable angina pectoris (Braunwald class 3)
* Patients with severe congestive heart failure
* Patients with severe heart failure NYHA IV
* Patients with severe valvular heart disease
* Women who are pregnant or lactating
* Patients with another coronary stent implanted previously into the target vessel, drug eluting stents less than 9 months and bare metal stents or stents with passive coatings less than 3 months before the PEPCAD IV DM PCI
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patients who had a cerebral stroke < 6 months prior to the procedure
* Patient participates in other clinical trials involving any investigational device or drug
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR<30ml/min) and is therefore not eligible for angiography. Patient's serum creatinine levels must be documented
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g., malignancy)
* Addiction to any drug or to alcohol
* Patients with any type of surgery during the week preceding the interventional procedure.
* Therapy with anticoagulants
* Poorly controlled diabetes mellitus as reflected by an HbA1c ≥ 8% during the six months prior to enrollment in PEPCAD IV DM
* Patient has a history of peptic ulcer or gastric/intestinal bleeding during the past 6 months.
* Evidence of extensive thrombosis within target vessel before the intervention
* Side branch > 2 mm in diameter originating from the lesion
* Stent within the same vessel less than 3 mm distant from target lesion
* Multi-lesion percutaneous coronary intervention within one vessel (PCI of a total of two lesions one each in a different vessels is permitted)
* Target lesion located in any type of coronary bypass (i.e., venous graft, arterial bypass) or graft/native artery connection
* Coronary artery occlusions of any type (e.g., acute or chronic)
* In-stent restenosis
* In-segment restenosis of the native vessel within 4 mm adjacent to the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-05; Primary Completion 2011-09 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Late lumen loss at 9 months | 9 months

SECONDARY OUTCOMES:
Procedural success | during procedure
Occurrence of acute (up to 48 hours), subacute (up to 30 days), and late thrombosis | 3 years
30-day MACE rate | 30 days
Percent in-stent stenosis at 9 months | 9 months
Percent in-segment stenosis at 9 months | 9 months
In-stent late loss index at 9 months | 9 months
Angiographic binary in-stent stenosis rate at 9 months | 9 months
In-segment late loss index at 9 months | 9 months
Angiographic binary in-segment stenosis rate at 9 months | 9 months
Acute and cumulative MACE rate at 9 months | 9 months
Cumulative MACE rate after 2 years | 2 years
Indication for premature follow-up | up to 9 months
Type of recurrence (Mehran-Classification) | 9 months
Target vessel failure | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosli M Ali, MD, Principal Investigator — Cardiology Department Institut Jantung Negara National Heart Institute
Locations (1):
- Cardiology Department, Institut Jantung Negara, Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Ali RM, Degenhardt R, Zambahari R, Tresukosol D, Ahmad WA, Kamar Hb, Kui-Hian S, Ong TK, bin Ismail O, bin Elis S, Udychalerm W, Ackermann H, Boxberger M, Unverdorben M. Paclitaxel-eluting balloon angioplasty and cobalt-chromium stents versus conventional angioplasty and paclitaxel-eluting stents in the treatment of native coronary artery stenoses in patients with diabetes mellitus. EuroIntervention. 2011 May;7 Suppl K:K83-92. doi: 10.4244/EIJV7SKA15. PMID 22027736